CLINICAL TRIAL: NCT00797121
Title: Effect of Preoperative Biliary Drainage on Postoperative Complications in Resectable Patients With Hilar Cholangiocarcinoma(Klatskin Tumor)
Brief Title: Preoperative Biliary Drainage for Resectable Hilar Cholangiocarcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Liang Li-jian, the First affiliated hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SUMS-5010; Cholangiocarcinoma; Surgery; Drainage
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Cholangiocarcinoma; Drainage; Surgery
Keywords: Cholangiocarcinoma; Drainage
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative biliary drainage (Experimental)
  Interventions: Procedure: Preoperative biliary drainage
- Controlled group (No Intervention)

INTERVENTIONS:
Procedure: Preoperative biliary drainage — Percutaneous transhepatic biliary drainage(PTBD) is performed under the guidance of ultrasound. The duration may be around four weeks to make the total bilirubin of patients lower than 85μmol/L.
  Arms: Preoperative biliary drainage

SUMMARY:
This study is to investigate whether preoperative biliary drainage can reduce the postoperative morbidity in patients with hilar cholangiocarcinoma.

DETAILED DESCRIPTION:
Preoperative biliary drainage(PBD) or not, is a Hot Spot issue in the management of Hilar cholangiocarcinoma. Surgeons from Japan tend to perform PTBD(Percutaneous Transhepatic Biliary Drainage) before a definite operation until the total bilirubin(TB) lower than 85μmol/L. For some patients needed to perform extended curative resection, PVE(Portal Vein Embolization) is performed and thus the duration of PBD may be around six weeks and the final TB is lower than 34μmol/L. Some tend to perform a definite curative operation in a short time after diagnosis. There is no RCT research on the effect of PBD for the resectable Hilar Cholangiocarcinoma patients to date.

ELIGIBILITY:
Inclusion Criteria:

* Patients newly diagnosed
* Resectable patients after imaging assessment and evaluation of general condition of the patient
* TB>85μmol/L
* WBC account more than 1.5×109/L, PLT account more than 100×109/L and HB account more than 100g/L
* No serious disease in heart, lung and kidney
* Written informed consent

Exclusion Criteria:

* Unresectable patients.
* Patients have received biliary drainage procedure such as PTBD before admission
* Complicated with chronic hepatitis
* Myocardia infarction record within six months
* Women in pregnancy
* Serious disease in heart, lung or kidney

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative complication | 30 days after operation

SECONDARY OUTCOMES:
Postoperative mortality | 30 days after operation
Overall survival, OS | May, 2013
Disease free survival, DFS | May, 2013

CONTACTS AND LOCATIONS:
Overall Officials: Lijian Liang, Study Chair — Department of hepatobiliary, the first affiliated hospital, Sun Yat-sen University; Xiaoyu Yin, MD, Principal Investigator — Department of Hepatobiliary, the first affiliated hospital, Sun Yat-sen University
Locations (1):
- Department of Hepatobiliary, the first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Jarnagin WR, Fong Y, DeMatteo RP, Gonen M, Burke EC, Bodniewicz BS J, Youssef BA M, Klimstra D, Blumgart LH. Staging, resectability, and outcome in 225 patients with hilar cholangiocarcinoma. Ann Surg. 2001 Oct;234(4):507-17; discussion 517-9. doi: 10.1097/00000658-200110000-00010. PMID 11573044
- [Background] Nimura Y, Kamiya J, Kondo S, Nagino M, Uesaka K, Oda K, Sano T, Yamamoto H, Hayakawa N. Aggressive preoperative management and extended surgery for hilar cholangiocarcinoma: Nagoya experience. J Hepatobiliary Pancreat Surg. 2000;7(2):155-62. doi: 10.1007/s005340050170. PMID 10982608